CLINICAL TRIAL: NCT00365014
Title: Analysis of Disease Progression for Aplastic Anemia, Myelodysplastic Syndrome, Acute Myeloid Leukemia and Benzene Poisoning in Shanghai, China.
Brief Title: Progression of Hematopoietic Diseases in Shanghai, China
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Fudan University (Other); University of Cincinnati (Other); ExxonMobil Biomedical Sciences, Inc. (Industry); British Petroleum P.L.C. (Industry); Chevron Corporation (Industry); ConocoPhillips (Industry); Exxon Mobil (Industry); Marathon Ashland (Unknown); Shell Chemicals (Industry)
Responsible Party: Sponsor
Other Study IDs: 02-0036
Record Dates: First submitted 2006-08-14; First posted 2006-08-16 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Hematologic Diseases
Keywords: aplastic anemia; myelodysplastic syndromes; cytopenias; acute myeloid leukemia; myelodysplastic/myeloproliferative diseases; benzene poisoning
MeSH Terms: conditions — Hematologic Diseases; Anemia, Aplastic; Myelodysplastic Syndromes; Cytopenia; Leukemia, Myeloid, Acute; Myelodysplastic-Myeloproliferative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Blood disease patients: People with blood diseases presenting at Shanghai hospitals

SUMMARY:
The purpose of this study is to identify and characterize blood diseases presenting at Shanghai hospitals and to compare them with respect to clinical presentation, phenotype, molecular characteristics, benzene or other exposures and genetic susceptibility.

DETAILED DESCRIPTION:
The purpose of this study is to identify and characterize blood diseases presenting at Shanghai hospitals and to compare them with respect to clinical presentation, phenotype, molecular characteristics, benzene or other exposures and genetic susceptibility. The format for these studies is a set of clinical series superimposed on a case-control design that enables integration of detailed clinical and molecular characterizations of disease pathogenesis together with an evaluation of potential confounding and interacting factors within a structured statistical analysis of benzene exposure.

ELIGIBILITY:
Inclusion Criteria:

Men and women 18 years or older Diagnosis of hematologic abnormality

Exclusion Criteria:

Children Non hematologic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with blood diseases
Sampling Method: Non-Probability Sample
Enrollment: 10757 (Actual)
Dates: Start 2003-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
blood diseases presenting at Shanghai hospitals | hospital stay
  characterization of people with blood diseases presenting at Shanghai hospitals

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Irons, PhD, Principal Investigator — University of Colorado at Denver and Health Sciences Ctr.
Locations (1):
- Joint Sino-US Clinical and Molecular Laboratory (JCML), Shanghai, China